CLINICAL TRIAL: NCT04444531
Title: Ozone Therapy for Patients With COVID-19 Pneumonia: Preliminary Report of a Prospective Case-control Study
Brief Title: Ozone Therapy and Coronavirus Disease of 2019 (COVID-19) Pneumonia
Status: Completed | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Marc Vives, Clinical Research Lead, MD, PhD, EDAIC, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Other Study IDs: COVID Networking group
Record Dates: First submitted 2020-06-22; First posted 2020-06-23 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ozone autohemotherapy plus standard treatment
- Standard treatment alone

SUMMARY:
The objective is to determine whether the use of ozone autohemotherapy is associated with a decrease in time to clinical improvement

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID-19 infection (diagnosed by nasopharyngeal swab performed on admission)
* severe pneumonia with baseline chest X-ray abnormalities;
* Oxygen saturation <94% on room air, and tachypnea with respiratory rate exceeding 30 per minute.
* Informed consent signed.

Exclusion Criteria:

* Not willing to participate in the study.

Age Groups: Child, Adult, Older Adult
Study Population: - Adults >18yo hospitalised patients confirmed COVID-19 infection (diagnosed by nasopharyngeal swab performed on admission), with severe pneumonia with baseline chest X-ray abnormalities + oxygen saturation <94% on room air, and tachypnea with respiratory rate exceeding 30 per minute.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | 28 days
  Clinical improvement was defined as a two-point reduction (relative to the patient's status on hospital admission) on a six-point ordinal scale, or discharge alive from the hospital, whichever came first. The six-point scale was as follows: death (6 points); extracorporeal membrane oxygenation or mechanical ventilation (5 points); noninvasive ventilation or high-flow oxygen therapy (4 points); oxygen therapy without need for high-flow oxygen or non-invasive ventilation (3 points); hospital admission without need for oxygen therapy (2 points); and discharged from hospital or reached discharge criteria (1 point). Discharge criteria were as evidence of clinical recovery (normalization of pyrexia, respiratory rate <24 per minute, oxygen saturation >94% on room air, and absence of cough) for at least 72 hours.

SECONDARY OUTCOMES:
Rate of patients with Clinical improvement at day 14 | 14 days
  Clinical improvement was defined as a two-point reduction (relative to the patient's status on hospital admission) on a six-point ordinal scale, or discharge alive from the hospital, whichever came first. The six-point scale was as follows: death (6 points); extracorporeal membrane oxygenation or mechanical ventilation (5 points); noninvasive ventilation or high-flow oxygen therapy (4 points); oxygen therapy without need for high-flow oxygen or non-invasive ventilation (3 points); hospital admission without need for oxygen therapy (2 points); and discharged from hospital or reached discharge criteria (1 point). Discharge criteria were as evidence of clinical recovery (normalization of pyrexia, respiratory rate <24 per minute, oxygen saturation >94% on room air, and absence of cough) for at least 72 hours.
Rate of patients with Clinical improvement at day 28 | 28 days
  Clinical improvement was defined as a two-point reduction (relative to the patient's status on hospital admission) on a six-point ordinal scale, or discharge alive from the hospital, whichever came first. The six-point scale was as follows: death (6 points); extracorporeal membrane oxygenation or mechanical ventilation (5 points); noninvasive ventilation or high-flow oxygen therapy (4 points); oxygen therapy without need for high-flow oxygen or non-invasive ventilation (3 points); hospital admission without need for oxygen therapy (2 points); and discharged from hospital or reached discharge criteria (1 point). Discharge criteria were as evidence of clinical recovery (normalization of pyrexia, respiratory rate <24 per minute, oxygen saturation >94% on room air, and absence of cough) for at least 72 hours.
Time to a 2-fold decrease of C-protein reactive from baseline | 28 days
Time to a 2-fold decrease of ferritin from baseline | 28 days
Time to a 2-fold decrease of Lactate Dehydrogenase from baseline | 28 days
Time to a 2-fold decrease of D-dimer from baseline | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinic Ibiza Hospital, Ibiza Town, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Hernandez A, Vinals M, Pablos A, Vilas F, Papadakos PJ, Wijeysundera DN, Bergese SD, Vives M. Ozone therapy for patients with COVID-19 pneumonia: Preliminary report of a prospective case-control study. Int Immunopharmacol. 2021 Jan;90:107261. doi: 10.1016/j.intimp.2020.107261. Epub 2020 Dec 5. PMID 33310665